CLINICAL TRIAL: NCT00148551
Title: Triamcinolone Acetonide as an Adjunctive Treatment to Verteporfin Therapy in Neovascular Age-Related Macular Degeneration: Randomized Placebo-Controlled Clinical Trial.
Brief Title: Triamcinolone Acetonide as an Adjunctive to VPDT in ARMD.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Canadian Retinal Trials Group (Other)
Collaborators: University of British Columbia (Other); QLT Inc. (Industry); Vancouver Hospital (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01 (C03 - 0236)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2007-07-30 (Estimated); Status verified 2007-07

CONDITIONS: Age-Related Macular Degeneration
Keywords: AMD; Triamcinolone; Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Triamcinolone Acetonide

INTERVENTIONS:
Drug: Triamcinolone Acetonide

SUMMARY:
A 24 - month Study looking at the the changes in visual acuity of patients receiving PDT therapy in conjunction with intravitreal triamcinolone.

DETAILED DESCRIPTION:
This study will evaluate the effect of Triamcinolone Acetonide in conjunction with photodynamic therapy for the treatment of sub-foveal choroidal neovascular membranes secondary to age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with predominantly classic, subfoveal CNV secondary to AMD.
* No previous PDT Treatment in study eye.

Exclusion Criteria:

* CNV from conditions, other than AMD.
* Other disease that could be responsible for decreased vision.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2004-01; Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
Changes in visual acuity from baseline.

SECONDARY OUTCOMES:
Change in lesion characteristics from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: David A Maberley, M.D., Study Director — University of British Columbia
Locations (1):
- Eye Care Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Maberley D; Canadian Retinal Trials Group. Photodynamic therapy and intravitreal triamcinolone for neovascular age-related macular degeneration: a randomized clinical trial. Ophthalmology. 2009 Nov;116(11):2149-57.e1. doi: 10.1016/j.ophtha.2009.04.032. Epub 2009 Sep 12. PMID 19748675